CLINICAL TRIAL: NCT05714176
Title: Comparative Clinical Study to Evaluate the Efficacy and Safety of Oral Liposomal Iron, Oral Iron Supported Lactoferrin and IV Iron Dextran in Children With Chronic Kidney Disease
Brief Title: Comparative Study Between Oral Liposomal Iron,Iron Supported Lactoferrin and IV Iron Dextran in CKD Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Salah El-Din, Critical care clinical pharmacist, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iron in CKD children
Record Dates: First submitted 2023-01-15; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: CKD - Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Lactoferrin; Iron-Dextran Complex

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liposomal iron (Experimental): 30 pediatric patients who will receive oral liposomal iron (Novoferr) 30 mg/day for 12 weeks.
  Interventions: Drug: Ferric Pyrophosphate Liposomal
- Iron supported Lactoferrin (Experimental): 30 pediatric patients who will receive oral iron supported Lactoferrin iron (Provan) 100 mg/day for 12 weeks.
  Interventions: Drug: Lactoferrin
- Iv iron dextran (Experimental): 30 pediatric patients who will receive IV iron dextran 50 mg/3 times weekly for 12 weeks.
  Interventions: Drug: Iron Dextran Injection

INTERVENTIONS:
Drug: Ferric Pyrophosphate Liposomal — 30 pediatric patients who will receive oral liposomal iron (Novoferr) 30 mg/day for 12 weeks.
  Other Names: Novoferr
  Arms: Liposomal iron
Drug: Lactoferrin — 30 pediatric patients who will receive oral iron supported Lactoferrin (Provan) 100 mg/day for 12 weeks.
  Other Names: Provan
  Arms: Iron supported Lactoferrin
Drug: Iron Dextran Injection — 30 pediatric patients who will receive IV iron dextran 50 mg /3 times weekly for 12 weeks.
  Arms: Iv iron dextran

SUMMARY:
This is a randomized, parallel study that will be conducted on pediatric patients with CKD.

DETAILED DESCRIPTION:
The study will be conducted on 90 pediatric patients with CKD who will be divided into 3 groups: Group l: 30 pediatric patients who will receive oral liposomal iron 30 mg/day for 12 weeks. Group 2: 30 pediatric patients who will receive oral iron supported iron 1 mg+ lactoferrin 100 mg/day for 12 weeks. Group 3: 30 pediatric patients who will receive IV iron dextran 50 mg/3 times weekly for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A) Pediatrics ≤18 year old male and female patients. B) Pediatrics with CKD stages 3-5.

Exclusion Criteria:

* A) CKD patients' ≥18 year old. B) Active bleeding C) Malignancy D) Anemia due to any disease other than CKD E) Blood Transfusions

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin measure | 3 months
  Measure oxygen in blood by measuring hemoglobin by coloremetric assay

SECONDARY OUTCOMES:
Biomarkers measure | 3 months
  changes in serum levels of biological biomarkers( measure IL-6, hepcidin and GDF-15 by ELISA assay).

CONTACTS AND LOCATIONS:
Overall Officials: Sahar K Hagazy, PhD, Study Chair — Tanta University; Mohamed SH Al-Haron, Study Chair — Menoufia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amanullah F, Malik AA, Zaidi Z. Chronic kidney disease causes and outcomes in children: Perspective from a LMIC setting. PLoS One. 2022 Jun 8;17(6):e0269632. doi: 10.1371/journal.pone.0269632. eCollection 2022. PMID 35675292
- [Background] Ammirati AL. Chronic Kidney Disease. Rev Assoc Med Bras (1992). 2020 Jan 13;66Suppl 1(Suppl 1):s03-s09. doi: 10.1590/1806-9282.66.S1.3. PMID 31939529
- [Background] Ueda N, Takasawa K. Role of Hepcidin-25 in Chronic Kidney Disease: Anemia and Beyond. Curr Med Chem. 2017;24(14):1417-1452. doi: 10.2174/0929867324666170316120538. PMID 28302014
- [Background] Moscheo C, Licciardello M, Samperi P, La Spina M, Di Cataldo A, Russo G. New Insights into Iron Deficiency Anemia in Children: A Practical Review. Metabolites. 2022 Mar 25;12(4):289. doi: 10.3390/metabo12040289. PMID 35448476
- [Background] Wojtaszek E, Glogowski T, Malyszko J. Iron and Chronic Kidney Disease: Still a Challenge. Front Med (Lausanne). 2020 Dec 18;7:565135. doi: 10.3389/fmed.2020.565135. eCollection 2020. PMID 33392212

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT05714176/Prot_SAP_000.pdf